CLINICAL TRIAL: NCT03656991
Title: Bikes For Life: Measuring the Effects of a Bicycle Distribution Program on Pediatric Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's Hospital Colorado (Other); UnitedHealthcare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-0344
Record Dates: First submitted 2018-08-23; First posted 2018-09-04 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: This is a stepped-wedge, randomized controlled trial. Possible subjects will be randomized to 1 of 4 groups. Each patient will serve as his or her own control. Within each stratum of four, patients will be randomly assigned to intervention initiation times (~130 per initiation time). Intervention initiation times will occur every other month up to a maximum of six months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0 month group (Experimental): Receive the bicycle intervention at 0 months after enrollment.
  Interventions: Other: Bicycle intervention
- 2 month group (Experimental): Receive the bicycle intervention at 2 months after enrollment.
  Interventions: Other: Bicycle intervention
- 4 month group (Experimental): Receive the bicycle intervention at 4 months after enrollment.
  Interventions: Other: Bicycle intervention
- 6 month group (Experimental): Receive the bicycle intervention at 6 months after enrollment.
  Interventions: Other: Bicycle intervention

INTERVENTIONS:
Other: Bicycle intervention

SUMMARY:
The investigators propose a study to evaluate the success of a bicycle distribution program in increasing physical activity level, decreasing sedentary activity levels and positively affecting body-mass index (BMI) in participants aged 6 to 12 years old with overweight or obesity, who do not already own a bicycle, and are patients at the Children's Hospital Colorado Child Health Clinic (CHC), Lifestyle Medicine Clinic, or Rocky Mountain Youth Clinics. The investigators anticipate that the receipt of a bicycle will increase physical activity level, decrease sedentary activity time and decrease or stabilize patients' BMI. The investigators will answer this research question by distributing bicycles to 525 children and conducting follow up visits over the course of a year to measure the outcomes of interest.

ELIGIBILITY:
Inclusion Criteria:

* Ages 6-12 years
* Do not own a bicycle
* BMI over 85% for age (overweight or obese)

Exclusion Criteria:

* Outside of state age range
* Not overweight or obese
* Already own a bicycle.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 525 (Actual)
Dates: Start 2012-04-06 (Actual); Primary Completion 2016-10-25 (Actual); Study Completion 2018-04-04 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index | Change from Baseline BMI through study completion up to 78 weeks
Change in Physical Activity | Change from Baseline Physical Activity through study completion up to 78 weeks
  Average time spent participating in physical activity
Change in Sedentary Activity | Change from Baseline Sedentary Activity through study completion up to 78 weeks
  Average time spent in sedentary activities

SECONDARY OUTCOMES:
Change in Consumption of sugary drinks | Change from Baseline Consumption of Sugary Drinks through study completion up to 78 weeks
  Number of sugary drinks consumed
Change in Consumption of Fast Food | Change from Baseline Consumption of Fast Food through study completion up to 78 weeks
  Number of times fast food was consumed
Change in Consumption of Fruits | Change from Baseline Consumption of Fruits through study completion up to 78 weeks
  Number of fruits consumed
Change in Consumption of Vegetables | Change from Baseline Consumption of Vegetables through study completion up to 78 weeks
  Number of vegetables consumed

CONTACTS AND LOCATIONS:
Overall Officials: Maya Bunik, MD, MSPH, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared outside of the study.